CLINICAL TRIAL: NCT01963923
Title: Effectiveness of a Preoperative Pulmonary Rehabilitation Program in Exercise Tolerance and Quality of Life in Patients Awaiting Lung Resection by Video-assisted Thoracic Surgery
Brief Title: Effectiveness of a Preoperative Pulmonary Rehabilitation Program in Patients Awaiting Lung Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Esther Gimenez Moolhuyzen, Physiotherapist, Hospital Juan Canalejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCP-RSG-2011
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: Pulmonary Rehabilitation; Lung Cancer Resection; Video-assisted thoracic surgery; Exercise tolerance; Quality of life
MeSH Terms: conditions — Lung Neoplasms | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation Group (Experimental): The rehabilitation group must complete at least 16 sessions of the Pulmonary Rehabilitation Program
  Interventions: Behavioral: Pulmonary Rehabilitation Program
- Control Group (No Intervention): The control group must complete only the outcome measures and continue with their clinical routine as specified by their physicians.

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation Program — The pulmonary rehabilitation program includes an endurance training with a cycloergometer, a strength training with elastic bands and two dairy sessions of incentive spirometry with a volume-oriented device.
  Other Names: Endurance training; Strenght training; Incentive Spirometry
  Arms: Rehabilitation Group

SUMMARY:
The purpose of this study is to establish the effectiveness of a preoperative pulmonary rehabilitation program in patients awaiting lung resection for lung cancer by Video-assisted thoracic surgery in order to improve exercise tolerance and quality of life. The investigators hypothesized that a pulmonary rehabilitation program including both endurance and strength training may improve exercise tolerance and quality of life measured with a submaximal exercise test and a quality of life questionnaire respectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis confirmed or suspected of lung cancer (either primary or metastatic)
* Be on the waiting list for lung resection by Video-assisted thoracic surgery
* Present at least one of the next conditions: Forced Expiratory Volume in 1 second (FEV1)<80% of predicted and/or Body Mass Index > 30 or/and >80 years old and/or two or more comorbidities (Arterial Hypertension, Chronic Obstructive Pulmonary Disease, Coronary Disease, Diabetes, Renal Failure and/or cancer.
* No smoking at the time of recruitment
* Signed Informed Consent

Exclusion Criteria:

* Chemotherapy or Radiotherapy in the previous 6 months before the Rehabilitation program.
* Thoracotomies or pneumonectomies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario A Coruña, A Coruña, Spain

REFERENCES:
- [Derived] Sebio Garcia R, Yanez-Brage MI, Gimenez Moolhuyzen E, Salorio Riobo M, Lista Paz A, Borro Mate JM. Preoperative exercise training prevents functional decline after lung resection surgery: a randomized, single-blind controlled trial. Clin Rehabil. 2017 Aug;31(8):1057-1067. doi: 10.1177/0269215516684179. Epub 2016 Dec 20. PMID 28730888

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the study period, 40 patients were recruited (20 per arm) but only 12 patients in the control group and 10 patients in the rehabilitation group were included in the analysis due to losses in follow-up
Period: 3 Weeks Post-surgery
Arm/Group | Control Group | Rehabilitation Group
Started | 20 | 20
Completed | 12 | 10
Not Completed | 8 | 10
Period: 3 Months Post-surgery
Arm/Group | Control Group | Rehabilitation Group
Started | 12 | 10
Completed | 10 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Rehabilitation Group | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.4) | 70.9 (6.1) | 70.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  Spain | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Exercise Tolerance
Description: Maximum time sustained (in seconds) during the constant-load cycle endurance test performed at 80% of the maximal workload achieved measured three weeks after hospital discharge in comparison with the control group.
Time Frame: Exercise tolerance 3 weeks after hospital discharge
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rehabilitation Group | Control Group
Number analyzed (Participants) | 10 | 12
Seconds | 459.7 (264.7) | 341 (216.3)

2. Primary Outcome: Exercise Tolerance
Description: Maximum time sustained (in seconds) during the constant-load cycle endurance test performed at 80% of the maximal workload achieved measured three months after hospital discharge in comparison with the control group.
Time Frame: Exercise tolerance 3 months after surgery
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rehabilitation Group | Control Group
Number analyzed (Participants) | 9 | 10
Seconds | 560.3 (273.3) | 271.5 (95)

3. Secondary Outcome: Health-Related Quality of Life
Description: Health-Related Quality of Life measured with the 36-Item Short-Form Health Survey Version 2 (SF-36) three weeks post-surgery. This scale is scored on a 0 - 100 scale, with higher scores referring to a better health-related quality of life. The scale compromises 8 subscales and two summaries (physial and mental).
Time Frame: Quality of life 3 weeks after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation Group | Control Group
Number analyzed (Participants) | 10 | 12
units on a scale | 38 (8.6) | 42.1 (8.4)

4. Secondary Outcome: Health-Related Quality of Life
Description: Health-Related Quality of Life measured with the 36-Item Short-Form Health Survey Version 2 (SF-36) three months post-surgery. This scale is scored on a 0 - 100 scale, with higher scores referring to a better health-related quality of life. The scale compromises 8 subscales and two summaries (physial and mental).
Time Frame: Quality of life post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation Group | Control Group
Number analyzed (Participants) | 9 | 10
units on a scale | 45.8 (5.8) | 44.7 (7.6)

5. Secondary Outcome: Upper Body Strength
Description: Upper body strength measured with the Arm-Curl Test of the Senior Fitness Test. The test measures the number of curl-arm movements with a 2.27kg or a 3.61 kg dumbbell for women and men respectively during 30 seconds.
Time Frame: 3 weeks post-surgery
Measure: Mean (Standard Deviation); unit: Repetitions
Groups:
- Control Group: Number of curl-up repetitions performed in 30" in the control group
- Rehabilitation Group: Number of curl-up repetitions performed in 30" in the rehabilitation group
Arm/Group | Control Group | Rehabilitation Group
Number analyzed (Participants) | 10 | 10
Repetitions | 17 (3.4) | 17 (3.2)

6. Secondary Outcome: Upper Body Strength
Description: as for outcome 5
Time Frame: 3 months post-surgery
Measure: Mean (Standard Deviation); unit: Repetitions
Groups:
- Control Group: Number of curl-up repetitions performed in 30" in the control group 3 months post-surgery
- Rehabilitation Group: Number of curl-up repetitions performed in 30" in the rehabilitation group 3 months post-surgery
Arm/Group | Control Group | Rehabilitation Group
Number analyzed (Participants) | 10 | 9
Repetitions | 16.1 (3.1) | 16 (3.1)

7. Secondary Outcome: Lower Body Strength
Description: Lower body strength measured with the sit-to-stand Test. The test consist of counting the number of full stands from a chair that can be completed in 30 seconds with arms folded across chest.
Time Frame: 3 weeks post-surgery
Measure: Mean (Standard Deviation); unit: Repetitions
Groups:
- Control Group: Number of sit-to-stand repetitions performed in 30" in the control group 3 weeks post-surgery
- Rehabilitation Group: Number of sit-to-stand repetitions performed in 30" in the rehabilitation group 3 weeks post-surgery
Arm/Group | Control Group | Rehabilitation Group
Number analyzed (Participants) | 10 | 10
Repetitions | 13.2 (5.86) | 12.2 (5.05)

8. Secondary Outcome: Lower Body Strength
Description: as for outcome 7
Time Frame: 3 months post-surgery
Measure: Mean (Standard Deviation); unit: Repetitions
Groups:
- Control Group: Number of sit-to-stand repetitions performed in 30" in the control group 3 months post-surgery
Arm/Group | Control Group | Rehabilitation Group
Number analyzed (Participants) | 10 | 9
Repetitions | 11.5 (2.55) | 14.9 (5.6)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Rehabilitation Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No